CLINICAL TRIAL: NCT03737500
Title: Standard Silicone-based Breast Implant vs. B-Lite® Light Weight Breast Implant for Reconstructive Surgery After Total Mastectomy and Post-Mastectomy Radiotherapy for Breast Cancer: a Randomized Clinical Trial
Brief Title: Standard Silicone-based vs. B-Lite® Light Weight Breast Implant After Total Mastectomy and Radiotherapy for Breast Cancer
Acronym: BLITE-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICS Maugeri - CE 2202
Record Dates: First submitted 2018-11-05; First posted 2018-11-09 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Breast Implant; Complications; Breast Implant Protrusion; Breast Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard silicone-based breast implant (Active Comparator): Participants candidated to total mastectomy and radiotherapy will receive immediate or delayed breast reconstruction by the use of standard silicone-based breast implant (i.e. the breast implant commonly used in our institution)
  Interventions: Device: Standard silicone-based breast implant
- B-Lite® light weight breast implant (Experimental): Participants candidated to total mastectomy and radiotherapy will receive immediate or delayed breast reconstruction by the use of B-Lite® light weight breast implant
  Interventions: Device: B-Lite® light weight breast implant

INTERVENTIONS:
Device: B-Lite® light weight breast implant — Definitive breast reconstruction after total mastectomy by the use of B-Lite® light weight breast implant
  Arms: B-Lite® light weight breast implant
Device: Standard silicone-based breast implant — Definitive breast reconstruction after total mastectomy by the use of silicone-based breast implants commonly used in our institution
  Arms: Standard silicone-based breast implant

SUMMARY:
Reconstructive surgery with breast implants after total mastectomy for breast cancer is invariably related to several possible complications, such as atrophy of surrounding tissues, skin thinning, capsular contracture, wound dehiscence and inframammary fold break. Such complications are promoted by elastic properties of tissues and their response to gravity forces exerted on breast implant weight, leading to microischaemic events. A poor cosmetic outcome may result up to breast implant exposure, and its removal may become necessary, thus compromising the quality of breast reconstruction. These complications are further favoured by post-mastectomy radiotherapy (PMRT), since irradiation could enhance microischaemia of peri-prosthetic soft tissues and muscle, with subsequent inadequate healing, fibrosis and thinning. Since PMRT has been associated to improved loco-regional control in node-positive breast cancer patients, its use has increased in recent years. On one hand, PMRT has improved loco-regional control but, on the other hand, it has increased the failure rate of breast reconstruction after total mastectomy. Change of timing in breast reconstruction (immediate vs. two-staged by use of tissue expander) has not decreased the complications rate after PMRT. Currently the failure rate of breast reconstruction after total mastectomy and PMRT ranges from 0% to 40%. The present study will recruit 80 participants affected by breast cancer candidated to total mastectomy with immediate breast reconstruction and subsequent PMRT or total mastectomy with reconstruction by tissue expander, subsequent PMRT and then definitive reconstruction with breast implant. Participants will be randomized in two experimental arms: 40 patients will receive final reconstruction by the use of standard silicone-based breast implant and the other 40 patients will receive B-Lite® light weight breast implant. Participants will be followed up at 1, 6, 12 and 24 months, and all patients will undergo breast MRI at 6 months. The primary goal of the present study is to evaluate the failure rate of breast reconstruction (i.e. the need of re-intervention for breast implant removal). Secondary end-points include the overall complications rate, MRI evaluation of breast implant and surrounding tissues, cosmetic outcomes and quality of life including participants' satisfaction with breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis with indication of total mastectomy and breast reconstruction
* Indication of post-mastectomy radiation therapy
* Availability to be followed up for 24 months
* Signature of informed consent

Exclusion Criteria:

* Patients candidated to breast-conserving surgery
* Contraindicated breast reconstruction (severe comorbidities, unfavourable survival outcome expected, distant metastases)
* Patients affected by other solid malignancies
* Pregnancy
* Participation to other clinical studies in the last three months

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Failure rate of breast reconstruction | 24 months
  Need of re-intervention for breast implant removal for any cause (such as breast implant exposure)

SECONDARY OUTCOMES:
Overall complications rate | 24 months
  Occurrence of any complication at any time point, such as: capsular contracture, wound dehiscence, skin/soft tissues necrosis, inframammary fold break, implant exposure treated conservatively, hematoma, peri-prosthetic fluid collection, wound/implant infection
Magnetic resonance imaging (MRI) of breast implant and surrounding tissues | 6 months
  MRI evaluation for skin/soft tissues thinning, capsular contracture, implant break, chronic seroma
Change in cosmetic outcome | 1, 6, 12, 24 months
  Objective evaluation of cosmetic outcome by jugular-nipple/areola complex (NAC) and NAC-inframammary fold distances to evaluate symmetry, objective evaluation of plastic surgeon with serial photographs
Change in Quality of life (QoL) measured with BIBCQ | 6, 12, 24 months
  QoL evaluation included patient's satisfaction with breast reconstruction using the Body Image after Breast Cancer Questionnaire (BIBCQ)
Change in Quality of life (QoL) measured with BREAST-Q | 6, 12, 24 months
  QoL evaluation included patient's satisfaction with breast reconstruction, using the BREAST-Q score

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Corsi, MD, Principal Investigator — Istituti Clinici Scientifici Maugeri Spa SB
Locations (1):
- Breast Unit - Istituti Clinici Scientifici Maugeri Spa SB, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Govrin-Yehudain J, Dvir H, Preise D, Govrin-Yehudain O, Govreen-Segal D. Lightweight breast implants: a novel solution for breast augmentation and reconstruction mammaplasty. Aesthet Surg J. 2015 Nov;35(8):965-71. doi: 10.1093/asj/sjv080. Epub 2015 Sep 1. PMID 26333989
- [Background] Christante D, Pommier SJ, Diggs BS, Samuelson BT, Truong A, Marquez C, Hansen J, Naik AM, Vetto JT, Pommier RF. Using complications associated with postmastectomy radiation and immediate breast reconstruction to improve surgical decision making. Arch Surg. 2010 Sep;145(9):873-8. doi: 10.1001/archsurg.2010.170. PMID 20855758
- [Background] Ascherman JA, Hanasono MM, Newman MI, Hughes DB. Implant reconstruction in breast cancer patients treated with radiation therapy. Plast Reconstr Surg. 2006 Feb;117(2):359-65. doi: 10.1097/01.prs.0000201478.64877.87. PMID 16462313
- [Background] EBCTCG (Early Breast Cancer Trialists' Collaborative Group); McGale P, Taylor C, Correa C, Cutter D, Duane F, Ewertz M, Gray R, Mannu G, Peto R, Whelan T, Wang Y, Wang Z, Darby S. Effect of radiotherapy after mastectomy and axillary surgery on 10-year recurrence and 20-year breast cancer mortality: meta-analysis of individual patient data for 8135 women in 22 randomised trials. Lancet. 2014 Jun 21;383(9935):2127-35. doi: 10.1016/S0140-6736(14)60488-8. Epub 2014 Mar 19. PMID 24656685
- [Background] Ho AY, Hu ZI, Mehrara BJ, Wilkins EG. Radiotherapy in the setting of breast reconstruction: types, techniques, and timing. Lancet Oncol. 2017 Dec;18(12):e742-e753. doi: 10.1016/S1470-2045(17)30617-4. PMID 29208440
- [Background] Baschnagel AM, Shah C, Wilkinson JB, Dekhne N, Arthur DW, Vicini FA. Failure rate and cosmesis of immediate tissue expander/implant breast reconstruction after postmastectomy irradiation. Clin Breast Cancer. 2012 Dec;12(6):428-32. doi: 10.1016/j.clbc.2012.09.001. Epub 2012 Oct 11. PMID 23062707
- [Background] Fowble B, Park C, Wang F, Peled A, Alvarado M, Ewing C, Esserman L, Foster R, Sbitany H, Hanlon A. Rates of Reconstruction Failure in Patients Undergoing Immediate Reconstruction With Tissue Expanders and/or Implants and Postmastectomy Radiation Therapy. Int J Radiat Oncol Biol Phys. 2015 Jul 1;92(3):634-41. doi: 10.1016/j.ijrobp.2015.02.031. Epub 2015 Apr 28. PMID 25936815